CLINICAL TRIAL: NCT05896033
Title: The Impact of Menthol Regulation for Cigarettes and E-cigarettes on Tobacco Use Patterns for Current Menthol Smokers
Brief Title: Impact of Cigarette and E-cigarette Menthol Regulation on Current Smokers of Menthol Cigarettes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Minnesota (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tracy Smith, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 00122898; 1R01DA055985-01A1 (NIH)
Record Dates: First submitted 2023-05-19; First posted 2023-06-09 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Smoking Prevention and Control
Keywords: Smoking; Menthol
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Menthol Spectrum Cigarettes and Menthol E-cigarettes (Experimental): Ppts will be randomly assigned to receive the menthol spectrum cigarettes and Njoy Ace menthol e-cigarettes. Will be used for the duration of the study (8 weeks) starting at the second visit.
  Interventions: Behavioral: Menthol Cigarettes; Behavioral: Menthol Flavored E-cigarettes
- Menthol Spectrum Cigarettes and Tobacco E-cigarettes (Experimental): Ppts will be randomly assigned to receive the menthol spectrum cigarettes and Njoy Ace tobacco e-cigarettes. Will be used for the duration of the study (8 weeks) starting at the second visit.
  Interventions: Behavioral: Tobacco Flavored E-cigarettes; Behavioral: Menthol Cigarettes
- Non-menthol Spectrum Cigarettes and Menthol E-cigarettes (Experimental): Ppts will be randomly assigned to receive the non-menthol spectrum cigarettes and Njoy Ace menthol e-cigarettes. Will be used for the duration of the study (8 weeks) starting at the second visit.
  Interventions: Behavioral: Non-Menthol Cigarettes; Behavioral: Menthol Flavored E-cigarettes
- Non-menthol Spectrum Cigarettes and Tobacco E-cigarettes (Experimental): Ppts will be randomly assigned to receive the non-menthol spectrum cigarettes and Njoy Ace tobacco e-cigarettes. Will be used for the duration of the study (8 weeks) starting at the second visit.
  Interventions: Behavioral: Non-Menthol Cigarettes; Behavioral: Tobacco Flavored E-cigarettes

INTERVENTIONS:
Behavioral: Non-Menthol Cigarettes — Ppts will be randomly assigned to a group that receives non-menthol cigarettes
  Arms: Non-menthol Spectrum Cigarettes and Menthol E-cigarettes; Non-menthol Spectrum Cigarettes and Tobacco E-cigarettes
Behavioral: Tobacco Flavored E-cigarettes — Ppts will be randomly assigned to a group that receives tobacco flavored e-cigarettes
  Arms: Menthol Spectrum Cigarettes and Tobacco E-cigarettes; Non-menthol Spectrum Cigarettes and Tobacco E-cigarettes
Behavioral: Menthol Cigarettes — Ppts will be randomly assigned to a group that receives menthol flavored cigarettes
  Arms: Menthol Spectrum Cigarettes and Menthol E-cigarettes; Menthol Spectrum Cigarettes and Tobacco E-cigarettes
Behavioral: Menthol Flavored E-cigarettes — Ppts will be randomly assigned to a group that receives menthol flavored e-cigarettes
  Arms: Menthol Spectrum Cigarettes and Menthol E-cigarettes; Non-menthol Spectrum Cigarettes and Menthol E-cigarettes

SUMMARY:
In a 2x2 design, current menthol smokers (N=240) will complete a baseline period before being assigned to a cigarette (menthol or non-menthol) and e-cigarette condition (menthol or tobacco-flavored e-liquid) and receiving a 7-week supply of cigarettes and e-cigarettes. The study builds upon our well-established methodology for simulating tobacco regulatory policies. To model a ban, smokers will be instructed to only use their assigned products. Primary outcomes include cigarette smoking and e-cigarette use during Week 6. However, because a menthol ban may impact the ability to abstain from smoking, the investigators will incentivize participants to abstain from smoking during Week 7 (continued e-cigarette use allowed) and assess the time to first lapse. Participants will complete daily electronic diaries assessing tobacco product use throughout, which will be corroborated by biomarkers for menthol, nicotine, and smoke. Finally, to maximize the utility of these data for FDA regulation, the investigators will assess whether any demographic or baseline smoking characteristics moderate the observed treatment effects, calibrate the treatment effects to the US adult menthol smoking population, and model the effects of menthol regulation in cigarettes and e-cigarettes on smoking and vaping-attributable deaths and life-years lost.

ELIGIBILITY:
Inclusion Criteria:

1. adults (21+) who a) have been smoking at least 5 cigarettes daily for one year
2. usual brand (the brand used most often) is mentholated
3. have a smartphone that can receive text messages and access the internet (necessary for diary completion).

Exclusion Criteria:

1. other tobacco and pharmacotherapy criteria
2. health and safety criteria
3. planning to move out of the area within the next 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in cigarettes per day | Week 1- Week 6
  Will be measured through week 6 of the study

SECONDARY OUTCOMES:
Fagerstrom Test for Nicotine Dependence | Week 1- Week 7
  Cigarette Dependence
Ability to abstain from smoking | Week 7
  Participants will complete a 1-week practice quit attempt in week 7; time to first smoking lapse will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No